CLINICAL TRIAL: NCT07103291
Title: The Effects of Isocapnic Respiratory Muscle Endurance Training on the Multidimensional Components and Neurophysiological Mechanisms of Exertional Breathlessness in Healthy Adults
Brief Title: Effects of Isocapnic Respiratory Muscle Endurance Training in Healthy Adults
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Collaborators: Mitacs (Industry)
Responsible Party: Principal Investigator, Jordan Guenette, Professor, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: H25-00744
Record Dates: First submitted 2025-07-10; First posted 2025-08-05 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-08

CONDITIONS: Healthy Adults
Keywords: Exercise physiology; Respiratory muscle training; Cycling; Competitive cyclists

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low frequency and intensity training (Sham Comparator): Participant will perform a respiratory training following a low intensity and frequency protocol
  Interventions: Other: Sham respiratory muscle endurance training
- Progressive high frequency and intensity training (Active Comparator): Participant will perform a respiratory training following a progressive intensity and frequency protocol
  Interventions: Other: Respiratory muscle endurance training

INTERVENTIONS:
Other: Respiratory muscle endurance training — Respiratory muscle endurance training program over 5 weeks.
  Arms: Progressive high frequency and intensity training
Other: Sham respiratory muscle endurance training — Respiratory muscle endurance training program over 5 weeks following a sham training procedure that is meant to elicit no physiologic changes.
  Arms: Low frequency and intensity training

SUMMARY:
Respiratory muscle training (RMT) strengthens breathing muscles and may improve exercise performance and reduce breathlessness. However, different training methods and devices create controversy in the field. Two main types of RMT exist: inspiratory muscle training (IMT) and respiratory endurance training, like voluntary isocapnic hyperpnea (VIH). While IMT is well-studied, the impact of VIH on breathlessness remains unclear. This study will use the Canadian-developed BreathWayBetter device to examine how 5 weeks of VIH affects breathing discomfort and muscle function. Findings may help personalize RMT for athletes and clinical patients, improving respiratory care and exercise tolerance.

DETAILED DESCRIPTION:
Purpose: to determine the effect of voluntary isocapnic hyperpnea (VIH) respiratory muscle training (RMT) using the BreathWayBetter training device on the multidimensional components of dyspnoea, as well as exercise performances measures.

Objectives and Hypothesis:

Objective 1: The first primary objective is to examine the effects of the BreathWayBetter (BWB) training device on the intensity and unpleasantness of dyspnoea during exercise, and to determine what sensory qualities of dyspnoea are primarily affected.

Hypothesis 1: Change in dyspnea intensity (pre vs post training) will be the same in the sham and training group, however, the reduction in dyspnea unpleasantness will be significantly greater in the training group. The training group will also have a greater reduction in breathlessness-related emotional ratings compared to the sham group.

Objective 2: The second primary objective is to examine the effects of the BreathWayBetter (BWB) training device on peak oxygen consumption (VO2peak) during the pre and post intervention incremental cycle exercise tests in both conditions.

Hypothesis 2: Change in VO2peak (pre vs post training) will be greater in the training group compared to sham group.

Objective 3: The secondary objective is to explore the relationship between exercise performance and the subjective perception of dyspnoea following training.

Hypothesis 3: The magnitude of change in exercise performance will be moderately correlated with the magnitude of change in dyspnoea in the training group.

Justification:

Respiratory muscle training (RMT) is a collection of techniques designed to enhance respiratory muscle function through improvements in strength and endurance. While several reviews state that RMT has been shown to improve exercise performance, respiratory muscle strength, and dyspnoea ratings, it remains a contentious field of research. This controversy may be driven, at least in part, due to the wide variation of training devices and protocols used throughout the literature. Two predominant forms of RMT are typically used in healthy adults, respiratory muscle strength training and respiratory muscle endurance training. The former, more commonly referred to as inspiratory muscle training (IMT), incorporates breathing against resistive loading, while the latter uses isocapnic hyperpnoea as a training stimulus.

Respiratory muscle endurance training in the form of voluntary isocapnic hyperpnea (VIH) requires individuals to perform purposeful breathing at a target frequency and depth to maintain over a set duration. In contrast to the high-force, and often unidirectional demands of respiratory strength training, VIH consists of low-force, high-velocity contractions of inspiratory and expiratory muscles, which may be more relevant breathing patterns for endurance sports such as running and cycling. However, previous research has largely focused on the use of IMT on sports performance and respiratory muscle strength. Interestingly, given the notable positive effect on respiratory muscle strength, the use of RMT to alleviate dyspnoea, or breathlessness has been poorly studied. Several studies have reported decreases in ratings of perceived breathlessness during exercise following IMT. However, these studies employed unidimensional measurements that capture only the overall severity of dyspnoea, lacking a qualitative assessment of its intensity, unpleasantness, or emotional response necessary for a comprehensive understanding of dyspnoea in response to VIH training.

While previous literature is sparse, several studies have suggested that reductions in perceptual ratings may provide insight into the etiology of the ergogenic effect of RMT. RMT may result in a delayed onset of respiratory muscle fatigue and subsequently attenuate the respiratory muscle metaboreflex at high intensities. This reflex reduces blood flow to the peripheral locomotor muscles in favour of redirection to the respiratory muscles. Therefore a reduction in competitive blood flow and improved lactate clearance may provide reasoning for the lower perceived exertion of the limb muscles and breathing discomfort ratings observed. It may be further suggested that reduced respiratory muscle fatigue stems from an improved aerobic capacity of the primary and accessory muscles due to RMT. Therefore, it is plausible that VIH RMT may reduce the energy cost of breathing and/or improve peripheral limb oxygenation, which subsequently may lessen the intensity and quality of exertional dyspnoea sensations. Lastly, VIH RMT may also lead to desensitization to continuous loading of the respiratory muscles and diminish the perception of dyspnoea, specifically in the affective dimension (i.e., unpleasantness and emotion).

There are no studies that have assessed the multidimensional components of dyspnoea following respiratory muscle endurance training (i.e., VIH) nor the physiological outcome measures that may be linked to improvements in the intensity and quality of dyspnoea. Accordingly, the investigators have designed a study that will perform a multidimensional analysis of dyspnoea to provide a more comprehensive understanding of the immediate perception and emotional response to VIH RMT.

The Isocapnic BreathWayBetter (Isocapnic Technologies Inc, Kelowna, Canada) is a commercially available, affordable, portable device, paired with the free user-friendly app that allows for personalized VIH training programs with visual guidance that can be performed anywhere. However, its efficacy in improving measures of perceptual responses, such as the distressing qualities of dyspnoea (e.g., unsatisfied inspiration) following a prolonged training regimen remains unknown. Therefore, the primary aim of this study is to investigate the effects of 5 weeks of respiratory endurance training with the BWB device on the multidimensional components of breathlessness.

Statistical analysis:

The normality of the data will be tested using the Shapiro-Wilk test. A two-way mixed analysis of variance (ANOVA) will be performed to assess whether there are significant differences in pre and post-test measures of Borg dyspnoea ratings and selected respiratory measurements at standardized exercise times. Additionally, this will assess if the changes from pre and post-intervention measures differ between the control and intervention groups. Peak exercise data (final 30 seconds) will be compared within groups with paired t-tests and between groups with independent t-tests. Spearman's correlation coefficients will be used to examine the association between change in exercise time and dyspnoea scores. In all cases, a P value < 0.05 will be considered statistically significant. All data will be presented as means ± standard deviation (SD).

ELIGIBILITY:
Inclusion Criteria:

* 18-55 years of age (inclusive)
* Male or Female (biological sex)
* Body mass index greater than 18 or less than 30 kg/m2
* Normal pulmonary function: FEV1/FVC > 0.70 and FEV1 ≥ 80%
* Able to read and understand English
* Regularly trains and/or competes at a regional, national, or international level as a road cyclist or triathlete
* Access to a device with the capability to download the Isocapnic app (Apple IOS or Google Play/Android) or the ability to use the Web Based application.

Exclusion Criteria:

* Currently smoke, vape, or use cannabis, or have a history of frequent smoking, vaping or cannabis use
* History of, or current symptoms of cardiopulmonary (i.e., lung and/or heart) disease (excluding controlled asthma)
* Heart problem; a serious infection within the body; a neuromuscular (nerve to muscle) or musculoskeletal (muscle, ligament and/or bone) disorder; or other health problem that will be made worse with exercise testing
* Contraindications to exercise testing defined as anything that would prevent exercise under proper and safe conditions (e.g. a problem with the heart or lungs, muscle or bone injury, a serious infection)
* Currently pregnant
* Required to read and understand English due to the nature of the consent form and study materials, including questionnaires and training instructions, which are only available in English.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Estimated)
Dates: Start 2025-08 (Estimated); Primary Completion 2026-08-01 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in dyspnoea ratings on the 0-10 Borg scale after respiratory endurance training | Up to 7 weeks
  Dyspnoea ratings on the 0-10 Borg scale will be recorded during and after incremental cardiopulmonary exercise testing on a stationary cycle ergometer. Dyspnoea ratings will then be compared between the pre- and post-intervention visits.
Difference in maximal oxygen consumption (VO2peak) following high intensity training program compared to sham comparator program. | Up to 7 weeks
  Changes in peak oxygen consumption (VO2peak) will be measured during an incremental cardiopulmonary exercise test on a stationary cycle ergometer and compared between intervention conditions.

SECONDARY OUTCOMES:
Correlation between changes from baseline in maximal oxygen consumption (VO2peak) and changes from baseline in dyspnoea ratings on the 0-10 Borg scale following respiratory endurance training. | Up to 7 weeks
  Peak oxygen consumption (VO2peak) in units of ml/kg/min and dyspnoea ratings measured on the 0-10 Borg scale will be measured during an incremental cardiopulmonary exercise test on a stationary cycle ergometer and compared between the pre- and post-intervention visits.

CONTACTS AND LOCATIONS:
Overall Officials: Jordan Guenette, PhD, Principal Investigator — University of British Columbia
Locations (1):
- St. Paul's Hospital, Vancouver, British Columbia, Canada